CLINICAL TRIAL: NCT01806038
Title: The Effect of Pharmacist-Provided Counseling Combined With Outpatient Dispensing at Hospital Discharge on the Incidence of Post-Discharge Drug-Related Problems and Healthcare Utilization
Brief Title: Drug-Related Problems and Healthcare Utilization Post-Hospital Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00042998
Record Dates: First submitted 2013-03-05; First posted 2013-03-07 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-04

CONDITIONS: Drug Related Problems Post Hospital Discharge; Healthcare Utilization; Discharge Medication Counseling
Keywords: Adverse events; Drug interactions; Healthcare utilization; Discharge medication counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RPh Counseling + Outpatient Dispensing (Experimental): On the day of discharge, a pharmacist will perform a chart review and medication reconciliation on all patients' discharge medications (for patients randomized to the intervention arm). Any medication discrepancies will be addressed with the patient's primary care team. At the time of discharge, the patient will receive his/her discharge medications dispensed from the Duke Outpatient Pharmacy, along with medication counseling by a licensed pharmacist.
  Interventions: Other: RPh Counseling + Outpatient Med Dispensing at Discharge
- Routine Med Dispensing + Counseling (Active Comparator): At hospital discharge, patients will receive standard discharge procedures and obtain discharge medications per their usual process
  Interventions: Other: Discharge Med Dispensing Plus Counseling - Current Practice

INTERVENTIONS:
Other: RPh Counseling + Outpatient Med Dispensing at Discharge — On the day of discharge, a pharmacist will perform a chart review and medication reconciliation on all patients' discharge medications (for patients randomized to the intervention arm). Any medication discrepancies will be addressed with the patient's primary care team. At the time of discharge, the patient will receive his/her discharge medications dispensed from the Duke Outpatient Pharmacy, along with medication counseling by a licensed pharmacist
  Arms: RPh Counseling + Outpatient Dispensing
Other: Discharge Med Dispensing Plus Counseling - Current Practice — At hospital discharge, patients will receive standard discharge procedures and obtain discharge medications per their usual process
  Arms: Routine Med Dispensing + Counseling

SUMMARY:
The goal of this study is to investigate whether pharmacist provided counseling and medication dispensing at the patient's bedside can provide better outcomes than the current discharge process at Duke University Hospital. This study will be single-site, prospective, randomized, cohort study. Patients who meet the inclusion and exclusion criteria, and provide consent will be included in this study.

DETAILED DESCRIPTION:
Two Adult General Medicine Services, which do not have a rounding pharmacist (RPh), will be identified by the investigators. Permission to approach the patients on each service will be obtained from the attending physician of each respective General Medicine Service at the beginning of each attending physician's time on service. The attending physician will be asked to communicate to the study personnel of situations in which patients should not be approached (i.e., patient has communicated disinterested in being approached about study participation opportunities and/or, in the opinion of the attending physician, the patient should not be approached).

Patients who will be recruited from pre-specified medical services will be screened for eligibility and, if deemed eligible, then will be approached by study personnel and asked if they would like to enroll in this study. If the patient accepts, written informed consent will be obtained and the patient will enter the study. Patients will be randomly assigned to either the intervention or control arm. Patients randomized to the intervention arm will receive discharge medications and pharmacist-provided discharge medication counseling prior to hospital discharge, and patients randomized to the control group will receive standard discharge procedures and obtain discharge medications per their usual process. After the patient has been enrolled in the study, study personnel will collect patient demographic data for study purposes, utilizing patient medical records and/or patient interviews. At discharge, patients will receive either the intervention or standard of care defined by the arm of the study to which each patient has been randomly assigned. After discharge, a maximum of seven attempts will be made via phone to contact all patients in both arms for follow up at 30 (+/- 7) days after discharge. During the follow phone call, a blinded pharmacist will conduct a structured interview to collect data for the study endpoints. The pharmacist conducting the interview will have the most recent discharge medication list (the list the patient received at his/her hospital discharge) from the patient's medication record to be used for comparison to the information gathered from the patient's interview 30 days post discharge.

Intervention Arm - After enrollment, a pharmacy technician not associated with the study will collect information necessary to process and fill the patient's discharge prescriptions by the Duke Outpatient Pharmacy. On the day of discharge, a pharmacist will perform a chart review and medication reconciliation on all patients' discharge medications (for patients randomized to the intervention arm). Any medication discrepancies will be addressed with the patient's primary care team. At the time of discharge, the patient will receive his/her discharge medications dispensed from the Duke Outpatient Pharmacy, along with medication counseling by a licensed pharmacist.

Control Arm - Patients will receive the standard discharge process provided by nurses and/or physicians. Patients will obtain outpatient medications per usual care.

Data Evaluation - After a patient has completed the phone follow up interview, two pharmacist co-investigators who have not been involved in the inpatient care of the patients will review the collected data to assess for adverse drug reactions and drug-drug interactions. When there is a disagreement between the pharmacists concerning the occurrence of an adverse reaction (including causality or severity), or a drug interaction (including severity), a third pharmacist co-investigator who was not involved in the inpatient care of the patient will review the patient's data to make a final decision concerning the disagreement. All patients who complete the follow up survey will be evaluated in this manner.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients age 18 years or older scheduled for discharge to self-care from a Duke University Hospital Adult General Medicine Service that does not have a rounding pharmacist
* Able to be contacted via phone within 30 days post-discharge
* Able to speak and understand English
* (For intervention patients) Have at least one prescription filled by Duke Outpatient Pharmacy and receive medication counseling by a pharmacist at the time of discharge
* Of sufficient physical or mental capacity to provide informed consent, understand the medication counseling, manage their own medications, and answer the telephone questionnaire

Exclusion Criteria:

* Patients receiving medication-related counseling from other pharmacists (e.g., transplant patients or new start warfarin patients) or other healthcare providers (e.g., diabetes educators) during their hospital stay and/or at time of hospital discharge
* Patients without a telephone for follow up
* Patients with hearing and/or visual impairment
* Patients discharged to police custody
* Patients who are likely to be discharged the same day as admission
* Patients who, in the judgment of the Attending Physician, are not candidates for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Drug-related problems (composite of adverse drug reactions, drug interactions, and failure to receive drugs) during the first 30 days post-hospital discharge | 30 days post-hospital discharge

SECONDARY OUTCOMES:
Healthcare utilization | 30 days post-hospital discharge
  Number of emergency department visits, urgent care visits, and unanticipated visits to outpatient providers
Hospital readmissions | 30 days post-hospital discharge
  Number of hospital readmissions
Treatment delays | Within 24 hours after hospital discharge
  Number of patients who experience treatment delays, defined as inability to obtain medications prescribed at discharge

CONTACTS AND LOCATIONS:
Overall Officials: Paul W. Bush, PharmD, MBA, Principal Investigator — Department of Pharmacy, Duke University Hospital
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States